CLINICAL TRIAL: NCT01653548
Title: Evaluating a Novel Method of Generalizing Emotion Regulation
Acronym: EMOGEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Pro00035922; 1R01MH095806-01A1 (NIH)
Record Dates: First submitted 2012-07-17; First posted 2012-07-31 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: Problems With Emotion Regulation; Psychological Distress; Difficulties Coping With Negative Emotions; Anxiety; Depression; Borderline Personality Disorder
Keywords: emotion dysregulation; borderline personality disorder; anxiety; depression; negative emotions; outpatient interventions for negative emotions; psychological distress; emotion regulation problems
MeSH Terms: conditions — Anxiety Disorders; Depression; Borderline Personality Disorder | interventions — Habituation, Psychophysiologic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- HR training + Portable HR (Experimental): 100 subjects who receive Habituation Reminder training and who have access to the HR via a cellular phone.
  Interventions: Behavioral: Habituation Reminder Training; Behavioral: Habituation Reminder; Behavioral: Habituation
- HR Training + no portable HR (Experimental): 50 subjects who receive Habituation Reminder training and who do not have access to the HR via a cellular phone.
  Interventions: Behavioral: Habituation Reminder Training; Behavioral: Habituation
- No HR training (Experimental): 50 subjects who do not receive HR training.
  Interventions: Behavioral: Habituation

INTERVENTIONS:
Behavioral: Habituation Reminder Training — Participants will hear a unique sound after habituating to a personal stressor.
  Arms: HR Training + no portable HR; HR training + Portable HR
Behavioral: Habituation Reminder — Participants will hear the habituation reminder outside of the lab via a cellular phone.
  Arms: HR training + Portable HR
Behavioral: Habituation — Participants will habituate to personally-relevant stressor.

SUMMARY:
The aim of the present project is to develop and evaluate a novel and brief method of generalizing habituation (i.e., calming down after being upset) from an original learning context in the laboratory to other contexts inside and outside the laboratory. Specifically, the primary aim of this project is to evaluate whether novel habituation reminders (HRs) introduced following personally-relevant emotional stressors reduce acute negative emotions and psychological distress outside of an original learning context. Using a team of basic and applied scientists, over 4 years the investigators expect to screen 420 adult outpatients to enroll 250 study participants who have extreme difficulties with emotion regulation. These 250 participants will be randomly assigned to one of eight experimental groups, with the experimental design leading them through 1 or 2 of 3 project experiments.

Actual enrollment: 372 adult outpatients signed consent and enrolled into the study. 222 participants were eligible and began the study. Out of the 222, 210 completed the study (as opposed to the desired 250).

Experiment 1 will evaluate whether novel auditory HRs following personally-relevant emotional stressors differentially reduce psychological distress and negative emotions (via self-report and psychophysiology), compared to no HRs, within the same and different lab contexts after a 1 week delay. Experiment 2 will evaluate whether HRs differentially reduce negative emotions, psychological distress, difficulties with emotion regulation, and psychiatric symptoms, compared to sham sounds outside the laboratory across a 1 week period, using 8x daily assessments of distress and emotions and automated HRs/shams when acute negative emotions are present. An automated server and cellular phone system will be used to assess distress and emotional states and to deliver HRs/shams. Experiment 3 will examine the feasibility, acceptability, and preliminary effect size estimates when participants self-initiate the use of HRs in their daily lives across a 2 week period when acute negative emotions are present. The specific randomization rules across the 8 groups are explained in detail in the full protocol .

Risks in this study may arise from 1) the assessment interviews and questionnaires, and 2) discussing and hearing self-reported distressing events. Initial analyses will focus on the success of randomization to groups. The investigators will examine group differences on possible covariates (e.g., demographic variables) and those that are different across conditions will be used as covariates. Preliminary analyses will examine distributional properties of primary outcome measures and correlations among outcome measures and possible covariates. The investigators will set alpha at .05 for all analyses of primary hypotheses. To examine the influence of psychiatric symptoms (compared to the HR) on primary outcomes, the investigators will examine the relationship between baseline clinically relevant psychiatric variables (e.g., symptom severity) and changes in SUDS, emotional arousal, and clinical outcomes over time and if appropriate include these variables in primary analyses. Full data analytic plans are described in the full protocol.

DETAILED DESCRIPTION:
Difficulties regulating emotional arousal in a skillful manner are common across many psychiatric disorders and may be central to some of the most severe and difficult-to-treat populations (e.g., borderline personality disorder). To immediately decrease negative affect, individuals who have difficulties regulating negative emotions often rely on maladaptive behaviors that are significant public health problems, including substance use, suicidal behavior, binging/purging, and other negatively reinforced behavior. Conventional approaches to generalization of emotion regulation skills outside the clinic (e.g., assigning therapy homework) are insufficient. New interventions are needed that directly and immediately reduce acute negative emotions and do not rely on patient compliance with homework assignments or other top-down approaches. Accordingly, the primary aim of this project is to evaluate whether novel habituation reminders (HRs) introduced following personally-relevant emotional stressors reduce acute negative emotions and psychological distress outside of an original learning context. Using a team of basic and applied scientists, over 4 years investigators will recruit 420 adult outpatients to enroll 250 participants who have extreme difficulties with emotion regulation to participate in 3 experiments.

Actual enrollment: 372 adult outpatients signed consent and enrolled into the study. 222 participants were eligible and began the study. Out of the 222, 210 completed the study (as opposed to the desired 250).

Before being recruited into the study, potential participants will complete a phone screen-a pre-experiment screening questionnaire or an online questionnaire to assess certain exclusion and inclusion criteria. Eligible participants will be invited to the study office to provide written informed consent and receive a clinical assessment, during which full inclusion and exclusion criteria will be assessed.

Using the method developed by Pitman and colleagues and used in studies of adults with PTSD, BPD, and other diagnoses, investigators will create four negative emotional arousal scripts that will be used in a random order during Exp. 1. In brief, the Clinical Assessor will ask the participant to describe five of the most recent (i.e., past two weeks) moderate stressors in their lives. Participants will write a description of each event, and the clinical assessor will work with the participant to establish a clear story for each event that can be recited in approximately 30 seconds. The assessor will then review the script, ask for any clarification, and then ask the participant to rank them from most to least stressful. Following the assessment, the clinical assessor or same sex experimenter will digitally record these scripts into .mp3 files, which will be used in random order as the emotional stressors in Exp. 1.

Experiment 1

-Design-In Exp. 1, the investigators will use a 2 (Learning Phase: HR v. No HR) X 2 (Testing Phase: Context same v. different) X 2 (Testing Phase: HR v. No HR) between-subjects factorial design.

Randomization-All participants will be randomized to condition, with oversampling for HR groups, by using an urn randomization procedure by the off-site study statistician. Urn randomization will be conducted using age and gender as matching variables.

Learning Phase (Day 1)Baseline-First, baseline subjective units of general psychological distress (SUDS; visual analogue scale from 0-100) and emotional arousal will be assessed using self-reported and psychophysiological (galvanic skin response) measures. The Study Coordinator will affix electrodes using standard procedures, and will use Biopac MP150 hardware and AcKnowledge software for data acquisition. The galvanic skin response device is not being tested for safety or efficacy in this study, and is not being used as a diagnostic device. Participants will complete a five-minute baseline, sitting in a comfortable chair quietly without sleeping in a temperature controlled, sound attenuated room. SUDS and self-reported baseline emotion (SAM) will be obtained at the end of baseline.

Next, the emotional stressor task will be administered to all participants by playing a stressful script which was created during the clinical assessment. Prior to hearing the script, participants will be instructed to listen carefully and to attempt to imagine the event as vividly as possible. The task proceeds as follows: (1) the stressor will be heard via headphones (30s), (2) participants are instructed via standardized instructions to imagine as vividly as possible the stressful experience (30s), (3) silence (30s), (3) self-report of emotional arousal and valence (SAM; 30s) will be obtained via a computer. This sequence will repeat a minimum of two and a maximum of four times, until habituation has occurred (return to mean baseline arousal). Habituation will be continuously monitored using a real-time monitoring program currently being used in the lab that samples arousal (GSR) every 500ms relative to the average baseline arousal. This method allows idiographic analyses of habituation to the stressor, and ensures that the HR is administered during habituation. Individuals who continue to have high levels of emotional arousal after completing the emotional stressor task will be asked to sit in silence for 10 more minutes (receiving the SAM every 120 seconds), and if habituation has yet to occur, they will be prompted to focus on their breath to help with relaxation for the next 10 minutes. Based on findings using this emotional stressor task suggesting that habituation occurs within 3 minutes for veterans with PTSD, the investigators are confident that the approach will result in habituation. Once habituation occurs, the HR will be heard via headphones 3 times (for a total of 6s) by participants randomized to hear the HR, whereas the No-HR participants will hear nothing.

The HR will be a series of neutral novel sounds lasting 6s, and will be the same series of sounds being used in current lab ongoing studies testing extinction reminders. After the HR is played, the Study Coordinator will use standardized instructions to tell participants to remember this sound as a reminder of calming down. Lastly, SUDS and self-reported emotional arousal measure will be assessed (SAM). Physiological data will be continuously measured throughout this period. Although it is not expected to occur frequently, data from participants who do not habituate will not be used in analyses, and additional participants run. After completing the stressor task, there will be a 15 minute break, followed by a second and third administration of the stressor task using the procedures outlined above, but with a different personalized stressor recording each time. Investigators will randomize the order of the recordings that the participants described during the clinical assessment. At the end of the third emotional stressor task, participants will be scheduled for their Testing Phase one week later.

Testing Phase (Day 2)-One week after the Learning Phase, participants will complete the Testing Phase for Exp. 1. Upon arrival, half of the participants will be randomly assigned to be tested in the original laboratory room from the Learning Phase (same room as Day 1) and the other half to a new room. In line with the investigators' previous learning studies using context manipulations, the new room in the Testing Phase will represent a very different context compared to the room from the Learning Phase. The novel testing room will have different size, lighting, and furniture. Using a scent machine, the novel room will have the smell of mint released during testing. In addition, to ensure that the experimenter does not function as a reminder of habituation from the Learning Phase, testing in the novel room will be done by a different experimenter than in the original Learning Phase. In both the original and novel testing rooms, the Testing Phase will begin with a baseline (same procedures as above). Next, a new recording of a personally relevant stressor will be played (same procedures as in Learning Phase). Participants in both rooms will be randomly assigned to hear the HR or hear nothing (No HR). The HR will be presented through headphones every 10 seconds after the onset of the stressor task. Measures of psychological distress and emotional arousal will be obtained (same procedures as in the Learning Phase). As in the Learning Phase, after 10 minutes or when habituation occurs as operationalized above, the stressor will end and self-reported psychological distress and emotional arousal will be assessed.

Experiment 2

-In both the original and novel testing rooms, the Testing Phase will begin with a baseline (same procedures as above). Next, a new recording of a personally relevant stressor will be played (same procedures as in Learning Phase). Participants in both rooms will be randomly assigned to hear the HR or hear nothing (No HR). The HR will be presented through headphones every 10 seconds after the onset of the stressor task. Measures of psychological distress and emotional arousal will be obtained (same procedures as in the Learning Phase). As in the Learning Phase, after 10 minutes or when habituation occurs as operationalized above, the stressor will end and self-reported psychological distress and emotional arousal will be assessed. Because groups 5 and 7 from Exp. 1 will have only heard the HR during the Testing Phase, and it may therefore be associated with the emotional stressor but not habituation, these participants will not be randomized into Exp. 2. The participants in Exp. 2 will be randomized to either hear the HR or a sham sound delivered via the automated server and cellular phone platform when negative emotions are endorsed. The result is a 2 (Day 1 HR v. No HR) X 2 (Phone HR v. sham sound) Latin square experimental design.

Procedure. At the conclusion of Exp. 1, the Clinical Assessor will orient participants to Exp. 2. Over the next week, participants receive eight calls each day (approximately one call every two waking hours), with each call lasting 1-2 minutes. For both experimental conditions (HR v. Sham), calls on the first day will be used to establish baseline levels of psychological distress (SUDS; 0-9), emotional valence (positive vs. negative; 1-9 scale; endpoints from the SAM used) and strength of emotional arousal (1-9; SAM), while no HRs will be delivered. On all other days, when participants report high emotional arousal (i.e., >4) and low valence (i.e., negative affect; <5), they will automatically hear the HR or sham sound based on randomization to Exp. 2 condition. The sham sound will be a series of neutral percussive sounds unrelated to the HR in form but equivalent on other relevant parameters (e.g., amplitude, length). After the HR or sham sound, all participants will provide self-reported psychological distress (SUDS) and emotional valence/arousal, in order to evaluate differential changes due to the HR or sham sound. After one week, participants will return to the laboratory to return the phone, receive compensation, and be debriefed. To further evaluate clinically meaningful changes due to the HR, the experimenter will collect pre-, and post-Exp. 2 assessments of symptoms of clinical outcome measures (e.g., symptoms of anxiety and depression When beginning Exp. 2, information will be given on how to use the phone (with hands-free headset), keep its battery charged, and how to call study staff. Phones will be restricted to study-related access and emergency numbers only. All calls will be conducted using a dedicated server and existing software in the lab. The software uses automated dialing and recorded prompts that ask participants to provide ratings on the phone keypad.

First, to mitigate the possibility that the phone will be stolen, sold, or not used, the Study Coordinator and participants will create a plan to use the phone. Second, self-report scales will be the same as those from Exp. 1. Third, calls will be during times that the patient will normally be awake. No participant identifying information will be accessible in the cell phone. All data from the phone are stored in real-time in a password-protected computer in the lab.

Experiment 3

-The primary aim of Exp. 3 is to evaluate the feasibility, acceptability, and preliminary effect size estimates of a self-initiated HR (n = 50. on psychological distress and acute negative emotions by hearing the HRs over two weeks. Investigators will examine: (1) frequency of calls in to hear the HR within and across participants at times in their daily life when they are having acute negative emotions, and (2) how laboratory HR training affects psychological distress and emotional arousal/valence in naturalistic settings over time.

Procedures. At the conclusion of Exp. 1, the Clinical Assessor will orient participants to Exp. 3. Participants will be asked to call the automated server during the next two weeks when they are feeling acute negative emotions. To facilitate use of the HR, the assessor will discuss expected upcoming stressful events, in particular those that occur daily or frequently, and explain how the phone can be used to cope with these stressful or emotionally arousing situations. Participants will also be told that they will receive three automated calls a day, beginning the next day. During the 2 week period, participants calling in to the lab will hear a brief greeting and an assessment of present SUDS, emotional arousal and valence. If the participant indicates emotional arousal >4 and valence < 5, the automated system will ask if they would like to hear the HR. If the participant does not meet these requirements or indicates that they do not want to hear the HR, they will instead hear a brief message thanking them for calling in. After the HR or thank you message, all participants will then be again asked to report SUDS, emotional arousal and valence, after which the call will end. The procedure for calls out will be identical to Exp. 2, except that all participants will receive 3 calls a day, have access to the HRs, and be able to choose whether to hear the HR. After two weeks, participants will return to the lab, give back the cell phone, complete an exit interview, and receive compensation.

Exp. 3 compliance enhancement strategies are the same as in Exp. 2, except for the incentive structure.

Interviews-Diagnostic exclusions and current/past prevalence of Axis I and II diagnoses will be determined by the Structured Clinical Interview for Mental Disorders-I and II. Intelligence Quotient (IQ) will be assessed with the Peabody Picture Vocabulary Test-Third Edition (PPVT-III). The Treatment History Interview (THI)will be used to assess previous and ongoing psychiatric services received. The THI will be administered at pre- and post-experiment time points. All interviews will be videotaped, and investigators will determine the reliability of every tenth interview. Exit interviews will be conducted at the end of Exp. 3 to assess participants' acceptability of the HR.

Physiological Measurement-Skin conductance will be measured using Ag-AgCl electrodes on the middle phalanx of the middle and ring fingers of the participant's non-dominant hand. The electrodes will be connected to a Biopac MP150 device in an adjacent room. Amplified signals of analog data are converted to digital form and filtered using Biopac's AcKnowledge Software, and are stored in a database on the computer.

Biochemical measures-Urinalyses (UA's) are conducted at diagnostic intake to rule out participants currently taking illicit or prescription substances known to affect psychophysiological arousal. The specimens will be screened on-site using the Biosite Triage Meter Plus.. Urine will be tested for cocaine, marijuana, opiates, methadone, amphetamines, barbiturates, and benzodiazepines. Results will be available within 30 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-55
* Currently receiving outpatient psychiatric treatment
* Elevated overall score on Difficulties with Emotion Regulation Scale (Mean DERS total score >= 90)
* Urine test negative for presence of substances (illicit substances; e.g., cocaine, opioids, methamphetamine, PCP, THC, Methadone). If urine test is positive for amphetamine, barbiturates and benzodiazepines and subjects take them as prescribed, these subjects are allowed.

Exclusion Criteria:

* Current mania
* Meets full criteria for any current psychotic disorder
* Currently/chronically homeless
* Current suicidal ideation with intent
* Psychiatric hospitalization within past 6 months
* Substance use disorder within past 6 months
* Unable to read, blind, or deaf
* PPVT < 70
* Suicide Attempt within past 6 months
* Not currently in outpatient psychiatric treatment (i.e. psychotherapy, medication management, etc)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 372 (Actual)
Dates: Start 2012-08; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Reduction in emotional arousal or speed to recovery from emotional arousal following a stressor. | baseline and week 1
  The investigators will examine psychophysiological and self-report measures of emotional stress.

SECONDARY OUTCOMES:
Phone use feasibility | weekly from week 1-week 3
  Feasibility will be assess by examining (1) frequency of calls to hear the HR, (2) changes in SUDS, emotional arousal/valence (Post-Pre), (3) change in daily emotional arousal assessed over time, and (4) change over time in clinical outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Mark Z Rosenthal, Ph.D., Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center-Civitan Bldg, Durham, North Carolina, United States

REFERENCES:
- [Background] Bradley R, Greene J, Russ E, Dutra L, Westen D. A multidimensional meta-analysis of psychotherapy for PTSD. Am J Psychiatry. 2005 Feb;162(2):214-27. doi: 10.1176/appi.ajp.162.2.214. PMID 15677582
- [Background] Collins BN, Brandon TH. Effects of extinction context and retrieval cues on alcohol cue reactivity among nonalcoholic drinkers. J Consult Clin Psychol. 2002 Apr;70(2):390-7. PMID 11952197
- [Background] Gratz, K. L. & Roemer, L. (2004). Multidimensional assessment of emotion regulation and dysregulation: Development, factor structure, and initial validation of the difficulties in emotion regulation scale. Journal of Psychopathology and Behavioral Assessment, 26, 41-54
- [Background] Milad MR, Pitman RK, Ellis CB, Gold AL, Shin LM, Lasko NB, Zeidan MA, Handwerger K, Orr SP, Rauch SL. Neurobiological basis of failure to recall extinction memory in posttraumatic stress disorder. Biol Psychiatry. 2009 Dec 15;66(12):1075-82. doi: 10.1016/j.biopsych.2009.06.026. Epub 2009 Sep 12. PMID 19748076
- [Background] Roth, A., & Fonagy, P. (2005). What works for whom? A critical review of psychotherapy research. New York, NY: Guilford
- [Background] Schmahl CG, Elzinga BM, Ebner UW, Simms T, Sanislow C, Vermetten E, McGlashan TH, Bremner JD. Psychophysiological reactivity to traumatic and abandonment scripts in borderline personality and posttraumatic stress disorders: a preliminary report. Psychiatry Res. 2004 Apr 15;126(1):33-42. doi: 10.1016/j.psychres.2004.01.005. PMID 15081625
- [Background] Stokes TF, Baer DM. An implicit technology of generalization. J Appl Behav Anal. 1977 Summer;10(2):349-67. doi: 10.1901/jaba.1977.10-349. PMID 16795561
- [Background] Hayes SC, Wilson KG, Gifford EV, Follette VM, Strosahl K. Experimental avoidance and behavioral disorders: a functional dimensional approach to diagnosis and treatment. J Consult Clin Psychol. 1996 Dec;64(6):1152-68. doi: 10.1037//0022-006x.64.6.1152. PMID 8991302
- [Background] Brooks DC, Bouton ME. A retrieval cue for extinction attenuates spontaneous recovery. J Exp Psychol Anim Behav Process. 1993 Jan;19(1):77-89. doi: 10.1037//0097-7403.19.1.77. PMID 8418218